CLINICAL TRIAL: NCT04557137
Title: Fatigue and Quality of Life in Patients With Neuroendocrine Neoplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Gitte Dam, MD, PhD, University of Aarhus
Other Study IDs: 1-10-72-1-20
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Neuroendocrine Tumors (NET) Health Related Qualito of Life (HRQoL)
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Somatostatin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- NET: Study A:
  A cross-sectional study that investigates 250 patients (Cohort A) with neuroendocrine neoplasia, encompassing both patients with neuroendocrine tumors (NET) and neuroendocrine carcinomas (NEC).
  Study B:
- Newly diagnosed NET: A prospective study that investigates 30 newly diagnosed NET patients over three months (Cohort B) who are offered palliative treatment with somatostatin analogues.
  Interventions: Drug: Somatostatin analog

INTERVENTIONS:
Drug: Somatostatin analog — 120 mg ipstyl every 28 days
  Groups: Newly diagnosed NET

SUMMARY:
Numerous studies describe HRQoL in other cancer types, whereas only sparse research has been done in NEN patients. We wish to investigate HRQol in NEN patients. Using a validated generic tool with normative values derived from a background population, allows us to compare the values healthy controls.

Methods

Study A:

A cross-sectional study that investigates 250 patients (Cohort A) with neuroendocrine neoplasia, encompassing both patients with neuroendocrine tumors (NET) and neuroendocrine carcinomas (NEC).

Study B:

A prospective study that investigates 30 newly diagnosed NET patients over three months (Cohort B) who are offered palliative treatment with somatostatin analogues.

DETAILED DESCRIPTION:
The diagnosis of cancer and living with cancer has an impact on patients' HRQoL. Numerous studies describe HRQoL in other cancer types, whereas only sparse research has been done in NEN patients.

Previous studies concerning the effect of cancer on HRQoL have been useful and help clinicians regulate treatment regimens in other cancer types. In advanced cancer patients, it is shown that Global QoL, physical, role, and emotional functioning improves during HPN and it wasin patients who are candidates for HPN according to the European guidelines.

Moreover, patients with laryngeal cancer who are offered partial or total laryngectomy experience a significant and fast decline in HRQoL compared to those who are offered transoral laser microsurgery. This study has improved clinician and patient decision-making.

Previous studies investigating HRQoL in NEN patients have methodological limitations; no reference groups, limited number of patients or including a heterogenos group of patietns. This lack of methodological quality may explain the inconsistency in the HRQoL results found in previous NEN studies.To our knowledge, only a few cross-sectional studies of larger patient groups compared to a background population have been published.

Both HRQoL and fatigue are likely to be affected in NEN patients. Using a validated generic tool with normative values derived from a background population, allows us to compare the values healthy controls.

Aim

* To quantify HRQoL and fatigue in a cross-sectional study (Study A) of a large group of patients with NEN
* To investigate the immediate effect of diagnosis and somatostatin-analogue treatment on new patients. A prospective study over the course of three months (Study B)
* To investigate the change in HRQoL and fatigue during follow-up. (a three year follow-up will be performed beyond this research year)

Hypothesis

* HRQoL will be significantly lower and fatigue significantly higher in NEN patients compared to the general population
* HRQoL will be significantly lower and fatigue significantly higher in NEC patients compared to NET patients.
* Newly diagnosed patients with NET starting somatostatin analogue treatment will improve their HRQoL and reduce fatigue after a follow-up period of three months.
* In patients with neuroendocrine neoplasia, HRQoL will remain unchanged in patients with stable disease and derease in patients with disease progression.

Methods

Study A:

A cross-sectional study that investigates 250 patients (Cohort A) with neuroendocrine neoplasia, encompassing both patients with neuroendocrine tumors (NET) and neuroendocrine carcinomas (NEC).

Study B:

A prospective study that investigates 30 newly diagnosed NET patients over three months (Cohort B) who are offered palliative treatment with somatostatin analogues.

ELIGIBILITY:
Inclusion Criteria: all newly diagnosed NET and NEC patietns Exclusion Criteria:None

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All newly diagnosed NET and NEC patients All patients will be recruited from the department of Hepatology and Gastroenterology and at the Department of Oncology, at Aarhus University Hospital. Inclusion will happen at standard follow-up visits for patients in Cohort A and at first visit/time of diagnosis and at three-month follow-up for patients in Cohort B. Inclusion time is expected to be 9-10 months.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
NET and NEC | 12 months
  HRQoL

CONTACTS AND LOCATIONS:
Locations (1):
- Gitte Dam, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: Undecided